CLINICAL TRIAL: NCT04854382
Title: Tailored Information About the Coronavirus for Patients With Chronic Kidney Disease
Acronym: TICCKD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ivar Anders Eide (Other)
Responsible Party: Sponsor-Investigator, Ivar Anders Eide, Consultant Doctor / Researcher, University Hospital, Akershus
Organization: University Hospital, Akershus (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REK 144084/2020
Record Dates: First submitted 2021-04-13; First posted 2021-04-22 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Digital health literacy; Health literacy; Fear of coronavirus; Self-perceived health; Teach-back
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Tailored information about coronavirus using information videos followed by a teach-back procedure
  Interventions: Behavioral: Tailored information
- Control group (No Intervention): Controls have access to information videos, but do not receive the teach-back procedure (the intervention)

INTERVENTIONS:
Behavioral: Tailored information — Tailored information about coronavirus for patients with chronic kidney disease by information videos followed by a teach back procedure
  Arms: Intervention group

SUMMARY:
Randomized clinical trial focusing on the effect of tailored information on Covid-19 for patients with chronic kidney disease stage 5 on health literacy, anxiety and self-perceived health.

DETAILED DESCRIPTION:
This single-center randomized open clinical trial in persons with chronic kidney disease stage 5 investigates the effect of information about coronavirus targeted at the study population, using study specific information videos followed by a teach-back method. We measure digital, functional, interactive and critical health literacy, fear of coronavirus and self-perceived health at baseline and end-of-study. Patients are followed from May-July 2021 through February 2022 (study period 7-9 months).

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease stage 5

Exclusion Criteria:

* Covid-19 during last 12 months. Dementia or other reason why cannot participate like major depression, psychosis or hospitalized persons with severe frailty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Digital health literacy | 9 months
  Digital health literacy measured by Electronic Health Literacy Scale (shortened eHEALS, Norman et al 2006), a questionnaire composed of 8 items measuring combined knowledge, comfort, and perceived skills at finding, evaluating, and applying electronic health information to health problems, Likert scale 1 (lowest, worst digital health literacy) - 5 (highest, best digital health literacy), with max score 40.

SECONDARY OUTCOMES:
Health literacy | 9 months
  Health literacy measured by Health Literacy Questionnaire (shortened HLQ, Osborne et al 2013), a questionnaire composed of 44 items (9 dimensions) measuring reading and writing skills (functional), interactive and critical literacy. Likert scale 1 (lowest, worst health literacy) - 4 (highest, best health literacy) for some items and 1 (lowest, similar) - 5 (highest) for other items with calculations of mean score for each of the 9 dimensions.
Self-perceived Health | 9 months
  Self-perceived health measured with the EQ-5D-5L (EuroQol Group 1990), a questionnaire composed of 5 items / dimensions (mobility, autonomy, daily activities, pain, and anxiety and depression), Likert scale 1 (lowest / best health) - 5 (highest / worst health) with max score 25
Anxiety / concern | 9 months
  Anxiety / concern measured by the questionnaire Fear of corona scale (Ahorsu et al 2020), Likert scale 1 (lowest, least concern) - 5 (highest, most concern) with max score 35

CONTACTS AND LOCATIONS:
Overall Officials: Ivar A Eide, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lørenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-11-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT04854382/Prot_000.pdf